CLINICAL TRIAL: NCT00297908
Title: Alcohol Based Hand Sanitizer: Can Frequent Use Cause an Elevated Blood Alcohol Level?
Status: Completed | Type: Observational
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Other Study IDs: C.2006.041
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2007-02

CONDITIONS: Healthy
Keywords: Ethanol levels; Dermal absorbtion

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Ethanol based hand sanitizers do not raise blood alcohol levels to a measurable amount. This study will determine to what extent, if any, heavy use of ABHS changes blood alcohol levels.

DETAILED DESCRIPTION:
Ethanol continues to be the most frequently abused intoxicant in the United States.4 Drug testing in various work environments has become commonplace during the past two decades and will at times include blood, breath, or urine alcohol testing.5 While valid reasons for false positive drug tests do occur, a plethora of unusual and dubious explanations have been likewise tendered. Medical Review Officers (MRO) involved in evaluating such reports rely on past case reports, knowledge of laboratory analytical techniques, and other scientific evidence to validate or negate claims of drug use in the workplace. ABHS are now found in most hospitals and health-care facilities.1,3 Only one human report of serum ethanol levels following frequent clinical use of the ABHS has been reported.7 This finding of a negative serum ethanol level in this case is likely to be reproducible in all clinical settings as the physician attempted to simulate the most extreme use of the product that would be consistent with labeling instructions. Since alcohol breathalyzer testing is based upon exhaled portions of ethanol found within the blood stream, this method of testing would likely be negative as well.

Participants will be the investigators and associate investigators of the study, who are all employees in the emergency department at Darnall Army Community Hospital. There will be no financial reward offered. Consent will be obtained on all participants. The study will be performed in the Darnall Emergency Department outside of regular duty hours. Enrolled subjects will apply 5 ml of the product (62% denatured ethanol alcohol manufactured by Kimberley-Clark) to both hands and rub until dry. This will be repeated 50 times over approximately 4 hours. Participants will have their blood drawn prior to, as well as, after completing the study. No other laboratory tests will be performed other than the alcohol level. Pre study blood alcohol levels will be ordered to assure a pre-study level of 0 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 50 years without liver or renal disease working in the emergency department to include residents and staff physicians.

Exclusion Criteria:

* Alcohol intake or exposure in the past 12 hours to include ABHS.
* Allergy to ABHS or any of its ingredients.
* Any rash on the extremities.
* Currently taking disulfiram , metronidazole, chloramphenicol, nitrofurantoin, tolbutamide, chlorpropamide, glyburide, glipizide, tolazamide, griseofulvin, chloral hydrate, acetohexamide, and third-generation cephalosporins.
* Liver or kidney disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5
Dates: Start 2006-02; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Michael Luszczak, DO, Study Chair — C.R.Darnall Army Medical Center
Locations (1):
- Darnall Army Community Hospital, Fort Hood, Texas, United States

REFERENCES:
- [Background] Hilburn J, Hammond BS, Fendler EJ, Groziak PA. Use of alcohol hand sanitizer as an infection control strategy in an acute care facility. Am J Infect Control. 2003 Apr;31(2):109-16. doi: 10.1067/mic.2003.15. PMID 12665745
- [Background] Meengs MR, Giles BK, Chisholm CD, Cordell WH, Nelson DR. Hand washing frequency in an emergency department. Ann Emerg Med. 1994 Jun;23(6):1307-12. doi: 10.1016/s0196-0644(94)70357-4. PMID 8198306
- [Background] Turner P, Saeed B, Kelsey MC. Dermal absorption of isopropyl alcohol from a commercial hand rub: implications for its use in hand decontamination. J Hosp Infect. 2004 Apr;56(4):287-90. doi: 10.1016/j.jhin.2004.01.005. PMID 15066739
- [Background] Compton WM, Conway KP, Stinson FS, Colliver JD, Grant BF. Prevalence, correlates, and comorbidity of DSM-IV antisocial personality syndromes and alcohol and specific drug use disorders in the United States: results from the national epidemiologic survey on alcohol and related conditions. J Clin Psychiatry. 2005 Jun;66(6):677-85. doi: 10.4088/jcp.v66n0602. PMID 15960559
- [Background] Smith DE, Glatt W, Tucker DE, Deutsch R, Seymour RB. Drug testing in the workplace: integrating medical review officer duties into occupational medicine. Occup Med. 2002 Jan-Mar;17(1):79-90, v. PMID 11726338
- [Background] Plouvier B, Lemoine X, De Coninck P, Baclet JL, Francois M. [Antabuse effect during the administration of a topical drug based on monosulfiram]. Nouv Presse Med. 1982 Oct 30;11(43):3209. No abstract available. French. PMID 7177842
- [Background] Miller MA, Rosin A, Crystal CS. Alcohol-based hand sanitizer: can frequent use cause an elevated blood alcohol level? Am J Infect Control. 2006 Apr;34(3):150-1. doi: 10.1016/j.ajic.2005.09.009. No abstract available. PMID 16630979